CLINICAL TRIAL: NCT00837304
Title: Colon Capsule Endoscopy Versus Standard Colonoscopy in Assessing Disease Activity in Patients With Ulcerative Colitis - A Prospective Trial
Brief Title: Colon Capsule Endoscopy Versus Standard Colonoscopy in Ulcerative Colitis
Status: Terminated | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: Med-B_CCE_vs_SC
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2009-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UC: Patients with known ulcerative colitis
  Interventions: Device: PillCam Colon Capsule; Procedure: Standard Colonoscopy

INTERVENTIONS:
Device: PillCam Colon Capsule — PillCam Colon Capsule: The PillCam Colon capsule has two cameras that enable the device to take video images from both ends. It is 31.11 mm in size and takes pictures at a rate of 4 frames per second. The delay mode allows recording of images from the esophagus and the stomach for 5 minutes before the capsule switches into sleep mode for 2 hours to save energy.
Procedure: Standard Colonoscopy — Standard Colonoscopy: Pts. undergo colonoscopy with a video colonoscope (CF H180 AI; Olympus, Tokyo, Japan).

SUMMARY:
The dimension of diagnostic procedures and therapy of chronic inflammatory bowel diseases largely depends on the degree of mucosal inflammation. Video colonoscopy is currently the gold standard in the evaluation of the mucosa in patients with Ulcerative Colitis (UC). PillCam Colon Capsule was developed by Given Imaging, Israel, as possible alternative imaging modality to evaluate mucosal changes in patients with UC. The colonic mucosa can be visualized and recorded by video while the colon capsule passes the colon.

Many patients suffering from UC ask their physician for possible alternative diagnostic imaging because they are uncomfortable with conventional colonoscopy.

The primary aim of the present study is to compare the new Pillcam Colon Capsule with standard colonoscopy with respect to assessing mucosal disease activity and localization of inflamed colonic mucosa in patients with known UC.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with
* known ulcerative colitis
* Indication for Standard Colonoscopy
* Informed Consent given by the patient

Exclusion Criteria:

* Patient has dysphagia
* Patient has congestive heart failure
* Patient has renal insufficiency
* Patient is known or is suspected to suffer from intestinal obstruction
* Patient has a cardiac pacemaker or other implanted electronical medical devices
* Patient is pregnant
* Patient has had prior abdominal surgery of the GI tract
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
a) disease activity of ulcerative colitis (modified Rachmilewitz score) b) extent of colonic manifestation of ulcerative colitis c) accuracy parameters (sensitivity, specificity) | 12 months

SECONDARY OUTCOMES:
a) patient comfort b) detection of polyps c) differences in recognition of disease activity (physicians, nurses) d) differences in findings in the group of physicians (inter-observer differences) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, MD, Principal Investigator — University of Muenster, Dept. of Medicine B
Locations (1):
- University of Muenster, Dept. of Medicine B, Münster, Germany